CLINICAL TRIAL: NCT03008941
Title: A Phase I/II Randomized, Double-Blind, Placebo Controlled Study of Repeated Low-Dose Fecal Microbiota Restoration in HIV-Infected Subjects. The REFRESH Study
Brief Title: Microbiota Restoration Therapy in HIV With Repeated Low-Dose Interventions
Acronym: REFRESH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Sergio Serrano-Villar, MD, PhD, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 165-16; GESIDA 9116 (Other: GESIDA Study group)
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: HIV Infection
Keywords: HIV; microbiota; inflammation; fecal microbiota restoration
MeSH Terms: conditions — HIV Infections; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT (Experimental): Fecal microbiota capsules (provided by Openbiome).
  Dosage:
  * Induction: 10 capsules (single dose)
  * Maintenance: 5 capsules, weekly, during 7 weeks.
  Interventions: Biological: FMT
- Placebo (Placebo Comparator): Placebo capsules (provided by Openbiome).
  Dosage:
  * Induction: 10 capsules (single dose)
  * Maintenance: 5 capsules, weekly, during 7 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FMT — Capsules with fecal microbiota from healthy donors
  Arms: FMT
Other: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
Altered interplay between gut mucosa and dysbiotic bacteria during HIV infection seems to contribute to chronic immune dysfunction. Manipulation of the intestinal microbiota with nutritional interventions exert limited immunologic effects, but a deep understanding of how these interventions could ameliorate gut dysbiosis and influence health among HIV-infected individuals remain unexplored. In this Phase I clinical trial, 30 HIV-infected subjects on effective ART with evidence of persistent immune dysfunction, indicated by a CD4/CD8 ratio<1 will be included and randomized to either repeated low-dose oral fecal microbiota transplantation or placebo during 8 weeks. The primary outcome will be safety. Secondary outcomes will include changes in CD4+ T cell counts, CD8+ T cell counts, CD4/CD8 ratio, inflammatory markers, T cell activation and markers of enterocyte barrier function through week 48. Engraftment on host microbiota will be examined using Illumina sequencing of the V3-V4 16S RNA, and changes in bacterial metabolism and in the plasma metabolite fingerprint will be studied by combination of untargeted mass spectrometry and two different and complementary separation techniques in bacterial and plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* On stable antiretroviral therapy with plasma HIV RNA <20 copies/mL during at least 48 weeks.
* CD4/CD8 ratio <1

Exclusion Criteria:

* Pregnancy
* Gastrointestinal diseases, including cirrhosis
* Active infections, including HCV
* EBV and/or CMV negative patients (donors are not screened for EBV/CMV).
* Planned used of chemotherapy or antibiotics
* Allergy to sodium chloride or glycerol (the former components are capsule ingredients Generally Recognized As Safe (GRAS)
* Current or planned use of antimicrobial agents (including prophylactic treatments against P. jiroveci) other than ART.
* Neutropenia <500 cells/uL or CD4 counts <350 cells/uL
* Patients unable to give informed consent
* Patients unable to comply with the protocol requirements
* Predicted death within time period of follow-up
* Any other condition for which the treating physician thinks the treatment may pose a health risk
* Dysphagia: oropharyngeal, esophageal, functional, neuromuscular (e.g. stroke, multiple sclerosis, ALS)
* History of aspiration
* History of gastroparesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From baseline through week 48

SECONDARY OUTCOMES:
Changes in CD4+ T cell counts | From baseline through week 48
Changes in CD8+ T cell counts | From baseline through week 48
  1. Inflammation: interleukin (IL)-6, high sensitivity C reactive protein (hs-CRP), interferon gamma-induced protein (IP)-10.
  2. Monocyte/macrophage activation: sCD14, SCD163,
  3. Gut epithelial integrity: zonulin-1, intestinal fatty acid binding protein (IFABP).
  4. Bacterial translocation: lipoteichoic acid (LTA)
  5. Indolamine deoxygenase-1 induction: kynurenine/tryptophan ratio
  6. Coagulation: D-dimers
Changes in CD4/CD8 ratio | From baseline through week 48
  1. Inflammation: interleukin (IL)-6, high sensitivity C reactive protein (hs-CRP), interferon gamma-induced protein (IP)-10.
  2. Monocyte/macrophage activation: sCD14, SCD163,
  3. Gut epithelial integrity: zonulin-1, intestinal fatty acid binding protein (IFABP).
  4. Bacterial translocation: lipoteichoic acid (LTA)
  5. Indolamine deoxygenase-1 induction: kynurenine/tryptophan ratio
  6. Coagulation: D-dimers
Changes in microbiota alpha diversity metrics | From baseline through week 48
Changes in microbiota Unifrac distances | From baseline through week 48
Changes in microbiota Canberra distances | From baseline through week 48
Changes in plasma Interleukin-6 levels | From baseline through week 48
Changes in plasma hs-CRP levels | From baseline through week 48
Changes in plasma lipoteichoic acid levels | From baseline through week 48
Changes in plasma LBP levels | From baseline through week 48
Changes in plasma kynurenine/tryptophan ratio | From baseline through week 48
Percentage of HLA-DR+/CD38+ T cells in blood | From baseline through week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Derived] Serrano-Villar S, Talavera-Rodriguez A, Gosalbes MJ, Madrid N, Perez-Molina JA, Elliott RJ, Navia B, Lanza VF, Vallejo A, Osman M, Dronda F, Budree S, Zamora J, Gutierrez C, Manzano M, Vivancos MJ, Ron R, Martinez-Sanz J, Herrera S, Ansa U, Moya A, Moreno S. Fecal microbiota transplantation in HIV: A pilot placebo-controlled study. Nat Commun. 2021 Feb 18;12(1):1139. doi: 10.1038/s41467-021-21472-1. PMID 33602945